CLINICAL TRIAL: NCT01869452
Title: Telephonic Platform of Follow up, Therapeutical Education and Coordination in Secondary Prevention in Patients With Heart Failure and Coronary Disease
Brief Title: Platform Therapeutic Education in Heart Failure and Coronary Disease
Acronym: METISCARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Resicard (Other)
Collaborators: union nationale de formation et d'evaluation en medecine cardio-vasculaire (Unknown)
Responsible Party: Principal Investigator, Pr Ariel Cohen, head of the departement of cardiology,Saint Antoine hospital , Paris, Resicard
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Platform
Record Dates: First submitted 2013-05-23; First posted 2013-06-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure; Acute Coronary Syndrome; Coronary Bypass Graft Stenosis of Native Artery Graft
Keywords: education; risk factors; quality of life; coronary disease; telephone follow up; dedicated nurse
MeSH Terms: conditions — Heart Failure; Acute Coronary Syndrome; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- therapeutic education class 1 (Other): patients in class 1 will have a follow up call with therapeutic education every 3 months. this is the light follow up.
  Interventions: Behavioral: therapeutic education
- therapeutic education class 2 (Other): patients in class 2 will have a follow up call with therapeutic education every month. this is the moderate follow up
  Interventions: Behavioral: therapeutic education
- therapeutic education class 3 (Other): patients in class 3 will have a follow up call with therapeutic education twice a month. this is the heavy follow up.
  Interventions: Behavioral: therapeutic education

INTERVENTIONS:
Behavioral: therapeutic education — knowledge of disease, risk factors, diet, medication, alert symptoms

SUMMARY:
A first therapeutic education is given before patient's discharge at the hospital, then a dedicated nurse follows patients through the phone,regularly according to patients' needs, continues to give advise on risk factors, information on medication and alert symptoms and therapeutic education.

DETAILED DESCRIPTION:
Patients are assigned to an arm accordingly to their needs: class 1 with light therapeutic education, class 2 with moderate education, class 3 with heavy education. Assignement is based on the first education diagnosis during hospitalization time.

Quality of life and patient's knowledge are regularly evaluated through questionnaires

ELIGIBILITY:
Inclusion Criteria:

* hospitalization for acute coronary syndrome (ST-segment elevation myocardial infarction ,no ST-segment elevation myocardial infarction ST , unstable angina)
* hospitalization for heart failure
* acute coronary syndrome < 3 months
* heart failure < 3 months
* coronary by-pass surgery < 3 months

Exclusion Criteria:

* complicated acute coronary syndrome (ventricular arrhythmia, heart failure, mechanical complications, cardiogenic shock)
* valvular cardiac pathology
* obstructive cardiomyopathy
* planned cardiac transplantation
* severe neurological or psychiatric troubles
* loss of autonomy
* other (refusal, language, nursing house, way of life not compatible with follow up, refusal of telephonic contacts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
number of patient with a better of quality of life | 1 year
  quality of life is evaluated with appropriate questionnaires

SECONDARY OUTCOMES:
number of patients who improve their knowledge of disease | 1 year
  Knowledge of disease includes risk factors, symptoms, medication, diet. It is evaluated with appropriate questionnaires.
number of hospitalizations during the follow up | 1 year
  hospitalizations are recorded during the year of follow up, with cause and duration.

CONTACTS AND LOCATIONS:
Overall Officials: ariel a cohen, md, Principal Investigator — Resicard
Locations (4):
- France (4):
  - Institut Coeur Effort Sante, Paris
  - Clinique Turin, Paris
  - Hopital Saint Antoine, Paris
  - Centre Cardiologique Alfred Kastler, Sarcelles